CLINICAL TRIAL: NCT00757939
Title: A Two-Part Cross-Sectional and Longitudinal Study to Assess Regional Cerebral Blood Flow by Dynamic Arterial Spin Labeling as an Alzheimer's Disease Biomarker as Compared to FDG-PET in Patients With Mild-to-Moderate Alzheimer's Disease and Cognitively Normal Elderly Subjects
Brief Title: A Study to Assess Regional Cerebral Blood Flow as an Alzheimer's Disease Biomarker Compared to Positron Emission Tomography in Patients With Mild-to-Moderate Alzheimer's Disease and Cognitively Normal Elderly Subjects (Study MK-0000-068)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0000-068; 2008_547
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease, MRI, PET
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AD Participants (Experimental): Participants with a diagnosis of mild-to-moderate AD
  Interventions: Other: MRI; Other: FDG-PET
- Cognitively Normal Elderly Participants (Experimental): Elderly participants with no cognitive impairment
  Interventions: Other: MRI; Other: FDG-PET

INTERVENTIONS:
Other: MRI — During the study all participants will have 4 total MRI scans: baseline, 1 week, 6 and 12 months.
Other: FDG-PET — 2 to 4 PET scans will be done over 12 months, 2 planned and 2 more if data from any of these are un-interpretable

SUMMARY:
The aim of the study is to determine if regional cerebral blood flow, measured by dynamic arterial spin labeling (dASL), can be a biomarker for stage of Alzheimer's disease. The study is designed to be conducted in 2 parts in participants with mild to moderate Alzheimer's disease, and participants with normal cognition. Various imaging studies will be done using magnetic resonance imaging (MRI) and positron emission tomography (PET) along with neurocognitive assessments. Participants who meet the study-entry criteria will have up to 8 study visits. Repeat imaging studies may be required if the initial data are incomplete or un-interpretable. The maximum number of PET scans during the study will be limited to four.

ELIGIBILITY:
Inclusion Criteria:

The prospective participant must meet, at least, all of the criteria below (among others determined by the study staff) to be eligible for study participation.

The participant:

* Has mild-to-moderate Alzheimer's Disease (AD), OR is considered cognitively normal;
* Has been on stable doses of any regularly used medications for 4 weeks prior to study start;
* Must have been on a stable dose for 12 weeks prior to study start, of any medications taken for AD.

Exclusion Criteria:

If the prospective participant meets any of the criteria below (among others determined by the study staff) they will NOT be eligible for study participation.

The participant:

* Is living in a nursing home or skilled nursing facility;
* Has severe AD;
* Cannot undergo MRI;
* Cannot undergo PET scans;
* Has a history of neurological or neurodegenerative disorders, other than AD within 2 years prior to study start;
* Has taken Tacrine or anti-parkinsonian medications within 3 months of study start;
* Has taken corticosteroids, blood thinners, narcotic analgesics, benzodiazepines, or certain antihistamines within 1 month of study start;
* Initiates, discontinues, or changes the dose of any AD treatment during the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Regional cerebral blood flow, as measured by dASL. | 1 week, 6 and 12 months
  Part I: regional cerebral blood flow, measured by dASL at Baseline and 1 week in AD participants and cognitively normal controls. Part II: regional cerebral blood flow, measured at 6 months and 12 months in AD participants and normal control participants.

SECONDARY OUTCOMES:
Rate of cerebral glucose consumption, MRglc, as measured by fludeoxyglucose-PET (FDG-PET) | 12 months
  Regional cerebral rate of glucose consumption, MRglc, as assessed by FDG-PET will be measured at Baseline in (Part I) and at 12 months in (Part II), in AD participants and normal control participants.
Resting state functional MRI blood-oxygen-level-dependent (fMRI BOLD) response | 1 week, 6 and 12 months
  The resting state fMRI BOLD (blood-oxygen-level-dependent) signal will be evaluated for 'Goodness-of-Fit' to the default mode network at Baseline, 1 week, and 6 and 12 months in AD participants and normal control participants.